CLINICAL TRIAL: NCT02793076
Title: Physical and Emotional Benefits of Group Dance Intervention for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Sciences in Philadelphia (Other)
Collaborators: Cancer Support Community of Greater Philadelphia (Unknown)
Responsible Party: Principal Investigator, Colleen Maher, Assistant Professor, University of the Sciences in Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 840697-4
Record Dates: First submitted 2016-05-23; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Cancer
Keywords: Posture; Body image; Dancing; Group; Survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bollywood Dance (Experimental): Bollywood dance is a routine that doubles as both physical and mental exercise.
  Interventions: Other: Bollywood Dance

INTERVENTIONS:
Other: Bollywood Dance — 8 week Bollywood Dance Program

SUMMARY:
The purpose of this mixed methods study is to evaluate the effects an 8-week group dance intervention can have on body image and posture in breast cancer survivors.

DETAILED DESCRIPTION:
The purpose of this mixed methods study is to evaluate the effects of an 8-week group dance intervention on body image and posture in breast cancer survivors.

Program Description: An 8-week dance intervention was held at a local cancer support center in the greater Philadelphia region. The study ran for 8 weeks, and each class was held once a week for 60 minutes. Every class consisted of a 5-10 minute stretching warm up leading to approximately 50 minutes of teaching light choreography set to Bollywood music.

Methods: This was a mixed methods study utilizing two quantitative assessments and a qualitative portion comprising of initial and exit surveys. Breast cancer survivors were recruited from a local non-profit cancer support community in the greater Philadelphia region. A sample of twelve women (n=12) fulfilled inclusion criteria of being diagnosed with and treated for breast cancer. Dropout rate was low, and only 1 person fit this criteria. Informed consent was sought after and obtained through the University of the Sciences in Philadelphia Institutional Review Board.

Procedure: Group dance intervention program lasted for 8 weeks in total with no control group. All twelve subjects participated in 60-minute dance sessions, once a week for 8 weeks. At the beginning and termination of this 8 week dance intervention, all subjects took a series of assessments including the Body Image Scale (BIS), postural assessment using the plumbline method, and initial and exit open-ended surveys to assess any additional benefits of the program.

Analysis: Data review was completed through Microsoft Excel and SOFA Statistics (version 1.4.6), a free statistical analysis program (available online for download at www.sofastatistics.com). Means and modes were found in demographics using Excel. Qualitative data was explored initially through reading surveys and noting repetitive points. Survey data was coded by highlighting and labeling segments of common responses to survey questions. To ensure findings were consistent, an independent reviewer was employed to verify coded data. Codes were later organized according to similarity to develop common themes. Themes found from initial and exit surveys were studied closer using a comparative analysis, to look for connecting themes from initial and exit surveys.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with and treated for breast cancer

Exclusion Criteria:

* Participants who attended less than 6 classes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Body Image Scale (BIS) | Day 1(at start of dance intervention) and 8 weeks (at conclusion of dance intervention
  BIS is a 10-item likert scale questionnaire developed to assess body image. In a study by Hopwood et al. (2001), the BIS showed high reliability (Cronbach's alpha=0.93) and good clinical and discriminant validity.
Change in Plumbline | Day 1(at start of dance intervention) and 8 weeks (at conclusion of dance intervention
  Photographs were taken from a lateral view to assess shoulder posture. After palpating for the acromion joint, a tape marker was placed on the mid-acromion process. Participants were asked to stand with feet hip distance apart and look straight ahead. A full body picture was then taken from the lateral profile view. Pages for Apple, a computer software available through Mac (versions 10.11.3 and higher) was used to place a digital plumbline marker, which was perpendicular to the lateral malleolus on each photo. A second digital line was placed perpendicular from the mid-acromion process to the plumbline marker. The horizontal distance from the mid-acromion process to the plumbline marker was measured (inches) for each photo.
Change in Qualitative Open Ended Surveys | Day 1(at start of dance intervention) and 8 weeks (at conclusion of dance intervention
  Initial and exit open-ended surveys to assess any additional benefits of the program

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Maher, OTD, Principal Investigator — University of the Sciences
Locations (1):
- Cancer Support Community, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No